CLINICAL TRIAL: NCT00507637
Title: Prospective, Open-label, Single-arm, Single-center Trial to Investigate the Tolerability of NT 201 and Quality of Life of Patients in the Treatment of Blepharospasm With Shortened Injection Intervals
Brief Title: Blepharospasm Short Interval
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: primary efficacy endpoint not attainable.
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRZ 60201-0703/1; 2007-000697-23 (EudraCT Number)
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Blepharospasm
MeSH Terms: conditions — Blepharospasm | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NT 201 (IncobotulinumtoxinA/Xeomin®) (Experimental)
  Interventions: Drug: NT 201

INTERVENTIONS:
Drug: NT 201 — Injection of up to 50 Units NT 201 (incobotulinumtoxinA/Xeomin®) per eye and injection visit (8 injections visits in total).
  Other Names: Xeomin®; IncobotulinumtoxinA; "Botulinum toxin type A (150 kiloDalton), free from complexing proteins"

SUMMARY:
The objective of this Phase II study is to show that pre-treated patients with BEB with the need of shortened injection intervals achieve an improved and stable quality of life level if they receive repeated NT 201 injections at short injection intervals. In addition, the tolerability of repeated shortened NT 201 administrations in patients with BEB including the development of neutralizing antibodies will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of bilateral BEB characterized by spontaneous, spasmodic, intermittent or persistent involuntary contractions of the orbicular oculi muscles
* Medical need for treatment with shortened injection intervals (< 12 weeks) confirmed by the patient and investigator
* Blepharospasm Disability Index (BSDI) at baseline visit before injection of > / = 1,6

Exclusion Criteria:

* Atypical variant of blepharospasm caused by inhibition of levator palpebrae muscle (apraxia of the eyelid)
* Generalized disorders of muscle activity (e.g. myasthenia gravis, Lambert-Eaton syndrome), as well as amyotrophic lateral sclerosis or any other significant neuromuscular disease which might interfere with the trial
* The previous three injections with Botulinum toxin Type A with more than 50 Units [U] per eye per injection session
* Treatment with Botulinum toxins for any indication other than BEB within 4 months prior to baseline and during the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The difference between the actual Blepharospasm Disability Index [BSDI] value at each follow up visit and the BSDI value at baseline. | From baseline up to week 62. Follow up visits include 8 injection visits (V2 to V8) with intervals of at least 6 weeks between injections.
  The BSDI includes 6 items to be assessed by a 5-point scoring (i.e., 0-4 points per item) ranging from "no impairment, "slight impairment", "moderate impairment", "severe impairment" to "no longer possible due to my illness". The 6 items are "Driving a vehicle", "Reading", "Watching TV", "Shopping", "Walking" and "Doing everyday activities".

SECONDARY OUTCOMES:
Change in Jankovic Rating Scale (JRS) score from baseline over time. | From baseline up to week 62
  The JRS ranges from 0-8 points and consists of the two items "Severity" and "Frequency" with five rating categories each (0-4 points).
Patient Evaluation of Global Response [PEGR] rated by patient at visits V2 to V8 and at follow-up visit | Week 6 up to week 62
  The PEGR scale is a descriptive subjective 9-point response self-rating scale ranging from "complete abolishment of signs and symptoms" (+4) down to "very marked worsening" (-4).

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Wabbels, MD, Principal Investigator — Universitaets Augenklinik Bonn
Locations (1):
- Universitaets Augenklinik, Bonn, Germany